CLINICAL TRIAL: NCT04729244
Title: Critical Review of Efficacy of Hemp Oil (CBD) Tincture and Cream for Treatment of Pain, Anxiety, Insomnia and Reduction of Opioid Use
Brief Title: The Study of Hemp Oil CBD for Evaluation of Efficacy and Safety in Treatment of Pain, Anxiety and Insomnia Management
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Advanced Pain and Rehab Specialists (Other)
Collaborators: Hemp synergistics (Unknown)
Responsible Party: Principal Investigator, Anuradha Anand, Medical Director/Physician, Advanced Pain and Rehab Specialists
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AA00001
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: CBD; Pain, Chronic; Anxiety; Insomnia; Opioid Use
MeSH Terms: conditions — Chronic Pain; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: One group will be taking CBD tincture, the other will be using CBD cream
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBD(hemp oil) cream (Active Comparator): cream 2000mg/1oz (50mg/dose) once daily dosing for a total of 4 weeks to area of most pain.Patients will record outcome in pain, anxiety, sleep, and report any adverse effects.
  Interventions: Drug: CBD
- CBD (Hemp oil) Tincture (Active Comparator): 1500mg CBD/30ml (50mg/dose) once daily dosing for total of 4 weeks. Patients will record outcome in pain, anxiety, sleep, and report any adverse effects.
  Interventions: Drug: CBD

INTERVENTIONS:
Drug: CBD — Hemp Oil
  Other Names: CBD tincture; CBD cream

SUMMARY:
The investigators are looking to conduct a study looking at the effects of cannabidiol (CBD) from Hemp Oil in patients with Chronic pain, anxiety and insomnia. It is believed that CBD will improve pain anxiety and sleep quality and reduce opioid use. The study will last a total of 4 weeks and involve onsite visits in addition to weekly pain assessments.

DETAILED DESCRIPTION:
The proposal is to conduct a interventional cohort pilot study to evaluate the effectiveness of CBD on the management of chronic pain, anxiety and insomnia.

Subjects will be pre-screened from new and existing patients as well as from referral sites for the diagnosis of chronic pain. Potential subjects will be screened for pain >3 months who are using oral analgesic including narcotics and or physical therapy to reduce pain.

Those meeting all inclusion and exclusion criteria will receive a comprehensive history and physical exam and undergo informed consented at the Screening Visit. Baseline survey data will be collected including various pain rating surveys. The patient's will be monitored for compliance to complete the weekly rating using a research phone application.

Subjects will receive either CBD tincture or CBD topical cream.This will be dosed daily for a total of 4 weeks. Patients will be evaluated on three pain rating scales: On initial evaluation and 4th week evaluation, patients will be asked to fill out The Brief Pain Inventory and Pain Disability Index. Once weekly, a Numeric Rating Scale.

On initial evaluation and at 4th week evaluation, narcotic dosing will be reviewed and recorded. Quality of sleep and anxiety scale will also be recorded for the four weeks using the Hamilton Anxiety scale and Sleep Quality Assessment at the start and end of the 4 weeks. At initiation and conclusion of study blood work to evaluated levels of CBD in each patient. Subjects will be screened for side effects as well as records of pain medication use throughout the duration of the study

ELIGIBILITY:
Inclusion criteria:

* Patients with pain >3 months who are using oral analgesic including narcotics and or physical therapy to reduce pain.
* Patient provides informed consent
* Older than 21 years old,
* Previously have used CBD or marijuana
* Speaks English

Exclusion criteria:

* Patients who are receiving interventional pain procedures or surgery within 30 days
* for their pain
* Patients who have had pain <3 months
* Presence of serious medical illness
* Pregnant females
* Use of P450 modifying medications.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain score | 4 weeks
  Pain will be reported weekly using the Numeric Rating Scale. On initial evaluation and 4 week evaluation, patients will be asked to fill out The Brief Pain Inventory and Pain Disability Index.
  The primary study endpoint will be compared between groups using the area under the curve.

SECONDARY OUTCOMES:
Anxiety score | 4 weeks
  Hamilton Anxiety scale will be used to assess change in anxiety score at the beginning and end of the study. The two scores will be used to assess any change in anxiety.
  Hamilton Anxiety Rating Scale (HAM-A) Assessment on 14 items on a scale of 0 to 4. Each item is scored on a scale of 0 (not present) to 4(severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. A higher score is a worse outcome.
Insomnia Score | 4 weeks
  Sleep Quality Assessment at the beginning and end of the study and the difference will be used to assess any change.
  Sleep Quality Assessment is based on The Pittsburgh Sleep Quality Index (PSQI), an effective clinical tool to assess sleep quality and efficiency.
  It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month.
  Scores for each question range from 0 to 3, with higher scores indicating more acute sleep disturbances The sum of the scores of the seven components is used to compute the global sleep quality score, ranging in value from 0 to 21. A score of 0 indicates no sleep difficulties, while more-severe sleep difficulties correspond to higher values for the global and component scores.
Narcotic use reduction | 4 weeks
  Using Prescription Drug Monitoring Program at the beginning and end of the study to asses any change in medication.
  The Prescription Drug Monitoring Program (PDMP) is an online database that houses prescribing and dispensing data for patients per state.
  It calculates MME. The total daily morphine milligram equivalents (MME) will be displayed on a patients profile.
  0 means no narcotic use and higher values show high narcotic use which is a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Pain and Rehab Specialists, Hermitage, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Age, sex, medical conditions
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 8 months after publication for 3 years
Access Criteria: researchers physicians will have access to the data upon request